CLINICAL TRIAL: NCT02956031
Title: Primary HPV Screening as an Indicator of Cervical Pre-invasive and Invasive Neoplasia in HIV-positive and -Negative Southern African Women
Brief Title: Screening Study for Cervical Pre-cancer and Cancer Prevention in South African Women.
Acronym: DiaVACCS
Status: Recruiting | Type: Observational
Sponsor: University of Pretoria (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Professor Greta Dreyer, Professor, University of Pretoria
Other Study IDs: DiaVACCS
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer; High Grade Sil; CIN2
Keywords: cancer prevention; cervical screening; cervical cancer; cervical disease; cervical neoplasm; HPV testing; immunocytochemistry; triage techniques
MeSH Terms: conditions — Uterine Cervical Neoplasms; Squamous Intraepithelial Lesions; Uterine Cervical Diseases | interventions — Mass Screening; Colposcopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV pos: those who serologically tested positive for HIV
  Interventions: Other: Screening; Other: Colposcopy; Procedure: LLETZ
- HIV neg: those who serologically tested negative for HIV
  Interventions: Other: Screening; Other: Colposcopy; Procedure: LLETZ
- HIV unk: those with no available serological test for HIV
  Interventions: Other: Screening; Other: Colposcopy; Procedure: LLETZ

INTERVENTIONS:
Other: Screening — Cervical specimen obtained using speculum examination and cervical collection bush.
Other: Colposcopy — Vaginal speculum examination followed by application of 2% acetic acid and lugol's iodine with inspection with colposcope and punch biopsies taken of abnormal areas.
Procedure: LLETZ — The above (see colposcopy) is followed by local anaesthetic with two dentist's ampoules of lignocaine and large loop excision using coagulation of the abnormal area (usually 2 x 3 x 1 cm).

SUMMARY:
Nearly 8 000 new cervical cancer cases are diagnosed in South Africa per year; many are still undiagnosed and about 50% of diagnosed cases succumb per year. Although the current prevalence of pre-cancer cervical disease is largely unknown, data from local studies suggest regional differences and an increase in the prevalence of cytological abnormalities when compared with historical data. Low frequency in cytology screening is the primary factor attributable to development of invasive cervical cancer and almost one-third of all cervical cancer patients had previous negative cytology. Due to the low sensitivity of cytology it can be assumed that the true prevalence of pre-cancer disease is underestimated by all available data. One round of optimal cervical cytology will detect around 50% of existing pre-cancer cervical disease as identified and proven using colposcopy and directed biopsy. It is now widely accepted that primary screening with a human papilloma virus (HPV) test can improve the sensitivity of screening and that even a single round of HPV screening can rapidly reduce the incidence of invasive cervical cancer and related mortality within a few years.

South Africa has a high prevalence of HIV infection and a delay in or failure to initiate antiretroviral therapy (ART). These facts, together with the largely unscreened status of the female population and the high incidence of cervical cancer all suggest that HPV infection and precursors to cervical cancer are both unusually common among South African women. Accurate current knowledge of the performance of newer generation HPV based screening tests in HIV-infected and general female population are essential for cost-analysis and planning for national prevention and screening programs. This study will aim to demonstrate the feasibility and efficacy of new generation HPV deoxyribonucleic acid (DNA) based screening assays in a South African setting.

The investigators hypothesize that HPV testing followed by normal and special cytology tests will be a successful screening model for a South African population.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent accepted and signed
* Health seeking behaviour or request for a cervical cancer screening test
* Willing and able to receive test result by automated text message or clinic visit

Exclusion Criteria:

* Current pregnancy
* Hysterectomy
* Current or previous treatment for gynaecological cancer
* Hesitant or unable to undergo screening and treatment if indicated

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a multicentric study carried out in South Africa. Women with unknown HIV status will be recruited from the general population, and HIV positive women from adult antiretroviral treatment (ART) clinics.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2038-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Number of women with histologically proven cervical intraepithelial neoplasia grade 2+ (CIN2+) detected using HPV DNA analysis with partial genotyping as primary screen test followed by cervical cytology and immunocytochemistry as triage tests | Detected on histology biopsy at colposcopy after initial HPV screening with simultaneous cytology and immunocytochemistry testing

SECONDARY OUTCOMES:
Number of women with CIN2+ detected using HPV DNA analysis with partial genotyping that is associated with HPV types 16, 18, 16 and/or 18, only other high risk types | Detected on histology biopsy at colposcopy after initial HPV screening with simultaneous cytology and immunocytochemistry testing

CONTACTS AND LOCATIONS:
Overall Officials: Greta D Dreyer, PhD, Principal Investigator — University of Pretoria
Locations (1):
- Steve Biko Academic Hospital, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Snyman LC, Richter KL, Lukhwareni A, Dreyer G, Botha MH, Van Der Merwe FH, Visser C, Dreyer G. Cytology compared with Hybrid Capture 2 human papilloma virus cervical cancer screening in HIV positive and HIV negative South African women. Int J Gynecol Cancer. 2023 May 1;33(5):669-675. doi: 10.1136/ijgc-2022-003897. PMID 36650011